CLINICAL TRIAL: NCT00137774
Title: A Phase II Study of Bevacizumab in Combination With Temozolomide in Patients With Advanced Neuroendocrine Tumors
Brief Title: Bevacizumab in Combination With Temozolomide in Patients With Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Genentech, Inc. (Industry); Schering-Plough (Industry)
Responsible Party: Principal Investigator, Matthew H. Kulke, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-272
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Neuroendocrine Tumors
Keywords: Metastatic Neuroendocrine Tumor; Advanced Neuroendocrine tumor; Bevacizumab; Temozolomide
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Bevacizumab; Temozolomide

INTERVENTIONS:
Drug: Bevacizumab — Given intravenously every other week. Participants can continue to receive study drug as long as there is no disease progression or serious side effects.
Drug: Temozolomide — Given once daily for one week followed by a one week rest period. This one-week on/one-week off scheduled will be continued as long as there is no disease progression or serious side effects.

SUMMARY:
The purpose of this study is to determine what effects (good and bad) bevacizumab and temozolomide have on patients with neuroendocrine tumors.

DETAILED DESCRIPTION:
Patients will receive temozolomide orally once daily for one week, followed by a one-week rest period. This one-week on/one week off schedule will continue for the duration of treatment unless significant side effects develop.

Bevacizumab will be administered intravenously every other week. After eight weeks (two cycles), a CT scan will be performed to see how treatment affected tumor growth.

Bactrim, an antibiotic, and acyclovir, an antiviral medicine, will be given in order to help prevent infection.

Blood tests will be done every other week to evaluate any side effects.

Once the study has been completed, a physical exam, vital signs, blood tests, and CT scan will be performed.

Patients will remain on the study as long as they continue to receive benefit from the treatment and there are no serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented locally unresectable or metastatic neuroendocrine tumor excluding small cell carcinoma
* Measurable disease > 1cm by spiral computed tomography (CT) or > 2cm by other radiographic technique
* ECOG performance status of 0-2
* Life expectancy of > 12 weeks
* Prior treatment with chemotherapy is allowed
* Total bilirubin < 2.0mg/dl
* AST < 5x upper limit of normal (ULN)
* Serum creatinine < 2.0mg/dl
* Absolute neutrophil count > 1,000/mm3
* Platelets > 100,000/mm3
* International Normalized Ratio (INR) < 1.5

Exclusion Criteria:

* Prior treatment with temozolomide, decarbazine or bevacizumab
* Clinically apparent central nervous system metastases or carcinomatous meningitis
* Clinically significant cardiovascular disease
* Major surgery, open biopsy, or significant traumatic injury within 28 days
* Pregnant or breast-feeding women
* Chronic, daily treatment with aspirin or nonsteroidal anti-inflammatory medication
* Serious, nonhealing wound, ulcer or bone fracture
* Evidence of bleeding diathesis or coagulopathy
* History of other disease or metabolic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-11; Primary Completion 2005-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To assess the response to bevacizumab in combination with temozolomide in patients with metastatic neuroendocrine tumors | 2 years

SECONDARY OUTCOMES:
To assess the time to progression, progression free survival and safety of bevacizumab in combination with temozolomide in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Matthew H. Kulke, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Insitute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Result] Chan JA, Stuart K, Earle CC, Clark JW, Bhargava P, Miksad R, Blaszkowsky L, Enzinger PC, Meyerhardt JA, Zheng H, Fuchs CS, Kulke MH. Prospective study of bevacizumab plus temozolomide in patients with advanced neuroendocrine tumors. J Clin Oncol. 2012 Aug 20;30(24):2963-8. doi: 10.1200/JCO.2011.40.3147. Epub 2012 Jul 9. PMID 22778320